CLINICAL TRIAL: NCT00486525
Title: Breast Cancer Survivors: Physical Activity, Inflammation, Fatigue, and Distress
Brief Title: Hatha Yoga in Improving Physical Activity, Inflammation, Fatigue, and Distress in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OSU-06137; NCI-2012-00564 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); R01CA126857 (NIH); NCT00526526 (obsolete NCT alias)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Depression; Fatigue; Pain
Keywords: fatigue; depression; pain; cancer survivor; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Pain; Breast Carcinoma In Situ | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Yoga Therapy (Experimental): Patients participate in a Hatha yoga session over 90 minutes twice weekly for 12 weeks. Patients are also encouraged to practice yoga at home using the appropriate DVD/video segments for the month.
  Interventions: Procedure: Yoga Therapy
- Arm II: Wait-List (No Intervention): Wait-listed women were told to continue performing their usual activities, and to refrain from beginning any yoga practice. After their final assessment they were offered the yoga classes.

INTERVENTIONS:
Procedure: Yoga Therapy — Patients will undergo yoga therapy
  Other Names: Yoga
  Arms: Arm I: Yoga Therapy

SUMMARY:
RATIONALE: Yoga may improve inflammation, fatigue, and depression in female breast cancer survivors.

PURPOSE: This randomized clinical trial is studying how well Hatha yoga works in improving physical activity, inflammation, fatigue, and distress in female breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the yoga intervention will decrease inflammation, fatigue, and depressive symptoms relative to the waiting-list controls in women who are stage 0-IIIa breast cancer survivors.

OUTLINE: Patients are stratified according to stage of cancer (stage 0 vs stage I vs stage II and stage IIIA) and prior radiation therapy (yes vs no). Patients are randomized to 1 of 2 intervention arms.

* Arm I (waiting-list control): Patients are encouraged to perform usual activities, but asked to refrain from any yoga practice or other related activities. After a six-month observation period, patients undergo yoga intervention as described in arm II .
* Arm II (yoga intervention): Patients participate in a Hatha yoga intervention session comprising body postures and breath control techniques for 1.5 hours twice a week for 12 weeks. Patients are encouraged to practice Hatha yoga at home. Patients complete daily diaries on home Hatha yoga practices and submit them at each session.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stage 0-IIIA breast cancer survivor
* Completed cancer treatment within the past 36 months (except for tamoxifen/aromatase inhibitors)

  * At least 2 months since prior surgery, adjuvant therapy, or radiotherapy, whichever occurred last
* Women who are not currently practicing yoga and have not participated in any of the following activities:

  * Meditation, tai chi, or related activities
  * Yoga or tai chi within the past 6 months
  * Had classes for or practiced yoga for more than 3 months
* Women who typically engage in a total of 5 or more hours of vigorous physical activity per week are not eligible
* No inflammatory breast cancer

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Hemoglobin ≥ 10 g/dL (patients with a hemoglobin of < 10 g/dL may be retested in 6 weeks after treatment of anemia and allowed to participate in study if blood counts recovered)
* Physically able to fully participate in yoga intervention

Exclusion criteria:

* Inability to comfortably get up and down from the floor 2-3 times in a session
* Breathing problems requiring use of oxygen
* Problems walking without a cane or walker assistance
* Prior knee or hip replacement with limited movement in the joint
* Inability to comfortably lie on the stomach
* Alcohol, or drug abuse
* Diagnosis of any of the following conditions:

  * Diabetes
  * Chronic obstructive pulmonary disease
  * Uncontrolled hypertension
  * Evidence of liver or kidney failure
  * Symptomatic ischemic heart disease
  * Significant visual or auditory problems
  * Mental disorder or cognitive impairment
  * Notable serious cardiovascular history (e.g., prior life-threatening abnormal heart rhythms)
  * Other medical conditions involving the immune system such as autoimmune and/or inflammatory diseases including rheumatoid arthritis and ulcerative colitis
* History of breast or any other cancer, except basal or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No regular use of medications with major immunological consequences (e.g., steroids)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-08; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Kiecolt-Glaser, PhD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Kiecolt-Glaser JK, Bennett JM, Andridge R, Peng J, Shapiro CL, Malarkey WB, Emery CF, Layman R, Mrozek EE, Glaser R. Yoga's impact on inflammation, mood, and fatigue in breast cancer survivors: a randomized controlled trial. J Clin Oncol. 2014 Apr 1;32(10):1040-9. doi: 10.1200/JCO.2013.51.8860. Epub 2014 Jan 27. PMID 24470004
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled a sample of 200 breast cancer survivors with respect to age, stage of cancer, and treatment modalities between October 2007 and April 2012 in the Ohio State University Medical Center. Women were recruited through oncologists' referrals, community print and web-based announcements, and breast cancer groups and events.
Pre-assignment Details: We assessed functional limitations during the screening session. Those who had mobility/functional limitations were dropped out before randomization.
Groups:
- Arm I: Yoga Therapy: Patients participated in a Hatha yoga session over 90 minutes twice weekly for 12 weeks. Patients were also encouraged to practice yoga at home. Patients recorded their total home/class practice time in weekly logs.
Period: Overall Study
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Started | 100 | 100
Completed | 94 | 87
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (9.8) | 51.3 (8.7) | 51.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 200
  Male | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 27.9 (5.3) | 27.6 (6.0) | 27.8 (5.7)
SAD [Mean (Standard Deviation); unit: cm] — Sagittal Abdominal Diameter
  cm | 20.7 (3.3) | 21.0 (3.6) | 20.8 (3.4)
Ethnicity [Number; unit: participants]
  Asian | 3 | 2 | 5
  Black or African American | 8 | 10 | 18
  White | 88 | 88 | 176
  Not Reported | 1 | 0 | 1
CES-D depressive symptoms [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiological Studies Depression Scale (CES-D) has been used extensively to measure depressive symptomatology. Each of the 20 items are rated on a four-point scale, yielding a total score that can range from 0 to 60. Higher values represent more depressive symptoms.
  units on a scale | 10.2 (8.2) | 11.2 (8.2) | 10.7 (8.2)
Usage of Cardiac Medication [Number; unit: participants] | 17 | 16 | 33
CHAMPS activity [Mean (Standard Deviation); unit: total hours/week] — The Community Health Activities Model Program for Seniors questionnaire (CHAMPS) assessed the weekly frequency and duration of various physical activities.
  total hours/week | 6.8 (6.3) | 5.8 (5.1) | 6.3 (5.7)
MFSI-SF Fatigue [Mean (Standard Deviation); unit: units on a scale] — The 30-item Multidimensional Fatigue Symptom Inventory-Short form (MFSI-SF) assesses behavioral, cognitive, physical, and affective expressions of fatigue. Items are rated on a 5-point scale indicating how true each statement was for the respondent during the last week (0=not at all; 4=extremely). The total score represents the sum of the subscales measuring general, physical, emotional, and mental fatigue, minus the vigor scale, providing a possible range of scores from -24 to 96, with higher scores indicating greater fatigue.
  units on a scale | 14.3 (19.6) | 17.3 (20.5) | 15.8 (20.1)
SF-36 Vitality [Mean (Standard Deviation); unit: units on a scale] — The SF-36's (RAND Health Survey) energy/fatigue (vitality) scale focuses on the frequency of feelings of fatigue over the last month. Standardized scores on the RAND SF-36 vigor/vitality scale range from 0-100, with higher scores indicating less fatigue.
  units on a scale | 48.6 (20.2) | 44.4 (20.9) | 46.5 (20.6)
Marital Status [Number; unit: participants]
  Single | 18 | 8 | 26
  Married | 68 | 72 | 140
  Separated/Divorced | 14 | 15 | 29
  Widowed | 0 | 5 | 5
Education level [Number; unit: participants]
  High School or Less | 5 | 7 | 12
  Some College | 27 | 22 | 49
  College Grad | 29 | 33 | 62
  Postgraduate | 39 | 38 | 77
Employment Status [Number; unit: participants]
  Employed full or part time | 71 | 66 | 137
  Unemployed | 15 | 20 | 35
  Retired | 14 | 14 | 28
Income level [Number; unit: participants]
  $0-$25,000 | 3 | 7 | 10
  $25,000-$50,000 | 18 | 15 | 33
  $50,000-$75,000 | 17 | 18 | 35
  $75,000-$100,000 | 23 | 23 | 46
  >$100,000 | 30 | 29 | 59
  No report | 9 | 8 | 17
Type of Treatment [Number; unit: participants]
  Surgery Only | 13 | 13 | 26
  Surgery + Radiation | 28 | 24 | 52
  Surgery + Chemotherapy | 23 | 23 | 46
  Surgery + Radiation + Chemotherapy | 36 | 40 | 76
Cancer Stage [Number; unit: participants]
  Stage 0 | 9 | 9 | 18
  Stage I | 46 | 43 | 89
  Stage IIA | 27 | 25 | 52
  Stage IIB | 10 | 13 | 23
  Stage IIIA | 8 | 10 | 18
HER2 Receptor Status [Number; unit: participants]
  Positive | 18 | 17 | 35
  Negative | 74 | 72 | 146
  Unknown | 8 | 11 | 19
Progesterone Receptor Status [Number; unit: participants]
  Positive | 73 | 69 | 142
  Negative | 23 | 26 | 49
  Unknown | 4 | 5 | 9
Estrogen Receptor Status [Number; unit: participants]
  Positive | 81 | 78 | 159
  Negative | 15 | 17 | 32
  Unknown | 4 | 5 | 9
Usage of Tamoxifen/Aromatase Inhibitors [Number; unit: participants] | 72 | 71 | 143
Post-menopausal [Number; unit: participants] | 76 | 77 | 153
Time since diagnosis [Mean (Standard Deviation); unit: months] | 16.3 (7.5) | 18.4 (8.5) | 17.3 (8.1)
Time since treatment [Mean (Standard Deviation); unit: months] | 9.9 (7.1) | 11.8 (8.5) | 10.9 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Stimulated ln (TNF-a)
Description: log-transformed Lipopolysaccharide (LPS) stimulated Tumor Necrosis Factor-alpha (TNF-alpha)
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: ln (pg/mL)
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 92 | 84
ln (pg/mL)
  Immediately post-treatment | 8.31 (0.041) | 8.39 (0.040)
  3 months post-treatment | 8.31 (0.042) | 8.44 (0.043)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Mixed effect models were used to test the intervention's effect on primary outcomes. Fixed effects included visit, intervention group, their interaction, and baseline outcome levels. Random effects included a subject-specific random intercept, accounting for within-subject correlation, and a random effect for yoga-group, accounting for the partially-nested data arising from small groups being present in the intervention arm but not in the control arm; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.075, 95% CI 2-sided [-0.19 to 0.039], Standard Error of Mean 0.058 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.25 to -0.015], Standard Error of Mean 0.06 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of ln (TNF-a) for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.021, 95% CI 2-sided [-0.060 to 0.018], Standard Error of Mean 0.02 — Model used continuous yoga practice frequency in place of group assignment to predict primary outcomes immediately post-treatment
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p = 0.063, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.038, 95% CI 2-sided [-0.079 to 0.0021], Standard Error of Mean 0.02 — Model used continuous yoga practice frequency in place of group assignment to predict primary outcomes 3 months post-treatment

2. Primary Outcome: Stimulated ln (IL-6)
Description: log-transformed Lipopolysaccharide (LPS) stimulated Interleukin-6 (IL-6)
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: ln (pg/mL)
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 92 | 84
ln (pg/mL)
  Immediately post-treatment | 9.68 (0.043) | 9.76 (0.044)
  3 months post-treatment | 9.69 (0.044) | 9.85 (0.047)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.079, 95% CI 2-sided [-0.2 to -0.042], Standard Error of Mean 0.062 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.28 to -0.031], Standard Error of Mean 0.064 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of ln (IL-6) for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.3, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.022, 95% CI 2-sided [-0.063 to 0.019], Standard Error of Mean 0.021 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.056, 95% CI 2-sided [-0.098 to -0.013], Standard Error of Mean 0.022 — [estimate comment as in outcome 1, analysis 4]

3. Primary Outcome: Stimulated ln (IL-1b)
Description: log-transformed Lipopolysaccharide (LPS) stimulated Interleukin-1 beta (IL-1b)
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: ln (pg/mL)
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 92 | 84
ln (pg/mL)
  Immediately post-treatment | 8.31 (0.077) | 8.42 (0.071)
  3 months post-treatment | 8.32 (0.079) | 8.55 (0.074)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.31 to 0.11], Standard Error of Mean 0.11 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.44 to -0.014], Standard Error of Mean 0.11 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of ln (IL-1b) for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.034, 95% CI 2-sided [-0.10 to 0.035], Standard Error of Mean 0.0235 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.078, 95% CI 2-sided [-0.15 to -0.0074], Standard Error of Mean 0.036 — [estimate comment as in outcome 1, analysis 4]

4. Primary Outcome: MFSI-SF Fatigue
Description: The 30-item Multidimensional Fatigue Symptom Inventory-Short form (MFSI-SF) assesses behavioral, cognitive, physical, and affective expressions of fatigue.
  Items are rated on a 5-point scale indicating how true each statement was for the respondent during the last week (0=not at all; 4=extremely). The total score represents the sum of the subscales measuring general, physical, emotional, and mental fatigue, minus the vigor scale, providing a possible range of scores from -24 to 96, with higher scores indicating greater fatigue.
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 96 | 90
units on a scale
  Immediately post-treatment | 6.1 (1.7) | 10.3 (1.4)
  3 months post-treatment | 5.4 (1.7) | 12.4 (1.4)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-8.5 to 0.15], Standard Error of Mean 2.2 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-11.4 to -2.7], Standard Error of Mean 2.2 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of MFSI-SF Fatigue for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.019, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -1.7, 95% CI 2-sided [-3.1 to -0.28], Standard Error of Mean 0.70 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -2.8, 95% CI 2-sided [-4.2 to -1.4], Standard Error of Mean 0.71 — [estimate comment as in outcome 1, analysis 4]

5. Primary Outcome: Vitality, SF-36
Description: The SF-36's (RAND Health Survey) energy/fatigue (vitality) scale focuses on the frequency of feelings of fatigue over the last month.
  Standardized scores on the RAND SF-36 vigor/vitality scale range from 0-100, with higher scores indicating less fatigue.
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 96 | 90
units on a scale
  Immediately post-treatment | 58.7 (1.9) | 52.3 (1.7)
  3 months post-treatment | 58.1 (1.9) | 51.6 (1.7)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [1.4 to 11.4], Standard Error of Mean 2.5 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [1.5 to 11.6], Standard Error of Mean 2.5 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of vitality (SF-36) for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = 2.1, 95% CI 2-sided [0.40 to 3.75], Standard Error of Mean 0.85 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = 2.5, 95% CI 2-sided [0.77 to 4.14], Standard Error of Mean 0.85 — [estimate comment as in outcome 1, analysis 4]

6. Primary Outcome: CES-D
Description: The Center for Epidemiological Studies Depression Scale (CES-D) is a self-report scale designed to measure current symptoms of depression rated on a four-point likert scale.
  Scores range from 0-60, with higher scores indicating a higher frequency of depressive symptoms.
Time Frame: Immediately post-treatment and 3 months post-treatment
Population: Any subjects who do not have any measurements post-baseline are excluded from analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Number analyzed (Participants) | 96 | 90
units on a scale
  Immediately post-treatment | 8.1 (0.69) | 9.2 (0.70)
  3 months post-treatment | 8.5 (0.69) | 9.7 (0.71)
Statistical Analysis 1: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.0 to 0.88], Standard Error of Mean 0.98 — Yoga minus Control immediately post-treatment
Statistical Analysis 2: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.2 to 0.69], Standard Error of Mean 0.99 — Yoga minus Control 3 months post-treatment
Statistical Analysis 3: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of CES-D for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.66, 95% CI 2-sided [-1.3 to 0.0039], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Arm I: Yoga Therapy vs Arm II: Wait-List; Secondary analysis on change of CESD for each 10 minute increase in yoga practice frequency, adjusting for baseline outcome levels, age, and SAD; Test type: Superiority or Other; p = 0.098, Mixed Models Analysis; The Kenward-Roger adjustment to the degrees of freedom was used to control Type I error rates; Slope = -0.56, 95% CI 2-sided [-1.2 to 0.10], Standard Error of Mean 0.34 — [estimate comment as in outcome 1, analysis 4]

ADVERSE EVENTS:
Time Frame: Post-intervention
Arm/Group | Arm I: Yoga Therapy | Arm II: Wait-List
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 2/100 | 0/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Yoga Therapy (N=100) | Arm II: Wait-List (N=100)
Recurrence of chronic back and/or shoulder problems (Musculoskeletal and connective tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
We did not compare yoga to an active control group; Fatigue and depressive symptoms were not used as part of the inclusion criteria. Accordingly, our data may underestimate yoga's potential benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes